CLINICAL TRIAL: NCT05960409
Title: Outcome of Chest Trauma Patients in One Year in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Abdelhameed, resident at cardiothoracic department, Sohag University
Other Study IDs: Soh-Med-23-07-06MS
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Chest Trauma Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- blunt chest trauma patients: patients with chest injuries due to a blunt trauma
  Interventions: Procedure: chest tube - emergency thoracotomy
- penetrating chest trauma patients: patients with chest injuries due to penetrating trauma
  Interventions: Procedure: chest tube - emergency thoracotomy
- polytraumatized patients: patients with multible traumas beside the chest injury
  Interventions: Procedure: chest tube - emergency thoracotomy
- chest trauma only patients: patients with only chest injuries
  Interventions: Procedure: chest tube - emergency thoracotomy

INTERVENTIONS:
Procedure: chest tube - emergency thoracotomy — chest tube is an inter-costal tube inserted intrathoracic in case of haemothorax and pneumothorax ,,,, emergency thoracotomy is an emergency exploration in severly injured patients

SUMMARY:
The history of chest trauma is as old as that of man himself. One of the earliest writings about chest trauma is found in the Edwin Smith Surgical Papyrus, written in 3000 bc.

Over the last century, there has been considerable reduction in the mortality of chest trauma owing to improved pre-operative care, availability of positive pressure ventilation, increasing availability of antibiotics, improvement of radiological techniques and improved lung toilets measures etc.

Chest trauma implies trauma to any or combination of different thoracic structures, which can be divided into 4 anatomical regions i.e. the chest wall, the pleural space, the lung parenchyma, and the mediastinum.

Trauma is one of the top ranking causes of accidental or unnatural deaths. Chest trauma is a significant source of morbidity and mortality worldwide. overall, it accounts for 25%-30% of all trauma related deaths and is implicated in an additional 25% of patients, who died from injuries.

In most cases, blunt chest trauma is by far the commonest and road traffic accidents account for 70%-80% of such injuries. Fire-arm injuries, falling from height, blast, stabs, and various acts of violence are the other causative mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* adults and children
* isolated chest trauma
* polytraumatized patients
* penetrating chest trauma
* blunt chest trauma

Exclusion Criteria:

* patients presented with cardiac arrest
* patients presented dead
* patients with glasco coma scale 5 or less
* patients with sever abdominal injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * males and females
  * adults and children
  * isolated chest trauma
  * polytraumatized patients
  * penetrating chest trauma
  * blunt chest trauma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
morbidity | 12 months
  Outcome will be defined as conservative management
mortality | 12 months
  Outcome will be defined as conservative management

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mommsen P, Zeckey C, Andruszkow H, Weidemann J, Fromke C, Puljic P, van Griensven M, Frink M, Krettek C, Hildebrand F. Comparison of different thoracic trauma scoring systems in regards to prediction of post-traumatic complications and outcome in blunt chest trauma. J Surg Res. 2012 Jul;176(1):239-47. doi: 10.1016/j.jss.2011.09.018. Epub 2011 Oct 5. PMID 22099585
- [Background] Grubmuller M, Kerschbaum M, Diepold E, Angerpointner K, Nerlich M, Ernstberger A. Severe thoracic trauma - still an independent predictor for death in multiple injured patients? Scand J Trauma Resusc Emerg Med. 2018 Jan 8;26(1):6. doi: 10.1186/s13049-017-0469-7. PMID 29310701
- [Background] Ekpe EE, Eyo C. Determinants of mortality in chest trauma patients. Niger J Surg. 2014 Jan;20(1):30-4. doi: 10.4103/1117-6806.127107. PMID 24665200
- [Background] Al-Koudmani I, Darwish B, Al-Kateb K, Taifour Y. Chest trauma experience over eleven-year period at al-mouassat university teaching hospital-Damascus: a retrospective review of 888 cases. J Cardiothorac Surg. 2012 Apr 19;7:35. doi: 10.1186/1749-8090-7-35. PMID 22515842